CLINICAL TRIAL: NCT02286830
Title: Magnolia Study Prolonged Protection From Bone Disease in Multiple Myeloma. An Open Label Phase 3 Multicenter International Randomised Trial
Brief Title: Prolonged Protection From Bone Disease in Multiple Myeloma
Acronym: Magnolia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Lund (Other)
Responsible Party: Sponsor-Investigator, Thomas Lund, MD Ph.D., Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMSG 22/14; 2014-001121-32 (EudraCT Number)
Record Dates: First submitted 2014-03-12; First posted 2014-11-10 (Estimated); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma
Keywords: osteolysis; zoledronic acid; osteonecrosis; bone markers; low-dose CT
MeSH Terms: conditions — Multiple Myeloma; Osteolysis; Osteonecrosis | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zoledronic acid (Active Comparator): treatment with zoledronic acid for 4 years
  Interventions: Drug: Zoledronic acid
- no treatment (Placebo Comparator): treatment with zoledronic acid withheld after two years
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid will be given to all participants for two years. Then patients will be randomized to A receive 2 more years of treatment or B stop treatment.
  Other Names: Zometa

SUMMARY:
Main hypothesis: Patients who continue zoledronic acid after year 2 have longer time until progression in bone disease compared to patients who stop treatment after two years?

Secondary hypothesis: Serum will bone markers increase prior to progression in bone disease in the individual patient?

Secondary hypothesis: Low-dose CT will detect more cases of osteolytic bone disease in Multiple Myeloma compared to conventional radiography

DETAILED DESCRIPTION:
Newly diagnosed myeloma patients will be followed for 4 years. The first two years they will be treated with zoledronic acid monthly. At year 2 they will be randomized to A continue treatment for 2 more years or B stop treatment. The primary outcome of the study will be time to progressive bone disease from year 2 and onward.

Serum bone markers will be measured throughout the study. In patients who experience progressive bone disease, development of bone markers prior to the radiological progression will be investigated to see the if it could have been predicted with the use of serum markers

During the four year period patients will have low-dose CT superior and conventional radiography made at predefined time points. The secondary outcome of the study is to compare the sensitivity of the two modalities

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Multiple Myeloma regardless of bone disease status
* Signed Informed Consent
* Age ≥ 18 years
* Remaining life expectancy ≥ 2 years
* Any concurrently anti-myeloma treatment are allowed

Exclusion Criteria:

* Previous treatment with bisphosphonate within the last 6 months
* Severely reduced renal function (creatinine clearance <30 mL/min despite fluid replacement)
* Known concurrent malignancy, excluding skin cancer
* Known hypersensitivity to zoledronic acid
* Pregnant or lactating women
* Women of childbearing potential or men engaging in sexual activity with a woman of childbearing potential who refuse to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
time to first skeletal related event after randomisations at year two | From year two to year four
  After two years of zoledronic acid treatment patients will be randomized to A continue treatment B stop treatment.

SECONDARY OUTCOMES:
Value of serum bone marker ratio (bone resorption / bone formation markers) as predictor of skeletal related related events analysed by time-dependent multiparameter Cox regression analysis. | 4 years
  Development in bone markers prior to progression in osteolytic lesions will be investigated

OTHER OUTCOMES:
Number of lesions identified with conventional radiography and low-dose CT | 4 years
  Patients will have low-dose CT and conventional x-ray made at predefined time points to compare the sensitivity between the two modalities
register incidence of osteonecrosis of the jaw | 4 years
register creatinine levels in serum | 4 years
  nephrotoxicity
register ionized calcium in serum | 4 years
  hypocalcemia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas LunD, MD Ph.D., Principal Investigator — Department of hematology, Odense University Hospital, Denmark
Locations (1):
- Odense University Hospital, Odense C, Denmark